CLINICAL TRIAL: NCT01220986
Title: An Observational Study of Liver Regeneration After Right Hepatectomy: Understanding the Molecular Primers of Liver Regeneration
Brief Title: Liver Regeneration After Liver Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: John S. Hammond, Division of Surgery, NIHR Nottingham Digestive Diseases Centre BRU
Other Study IDs: NDDC10/H0403/32
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Liver Diseases; Hepatectomy
Keywords: Liver regeneration; Innate immune response
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver tissue & serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Right hepatectomy: Intervals from inflow division.
  Interventions: Procedure: Liver biopsy

INTERVENTIONS:
Procedure: Liver biopsy — 0, 30, 60, 90 min post inflow-division

SUMMARY:
The aim of this study is to characterize Kupffer cell activity and activation of the innate immune response in the early phase of liver regeneration after right hepatectomy. The investigators hypothesise that liver regeneration after right hepatectomy in humans is associated with Kupffer cell activation and initiation of the innate immune response and that impaired liver regeneration, liver failure and sepsis following liver resection are associated with Kupffer cell dysfunction and an impaired innate immune response. The objectives for this study are to characterise Kupffer cell activity and the innate immune response in human liver before and after right hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring right hepatectomy for colorectal liver metastases

Exclusion Criteria:

* Age >75, neoadjuvant chemotherapy, recurrent disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing right hepatectomy for colorectal liver metastases.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dileep N. Lobo, DM FRCS, Study Chair — Reader in Surgery
Locations (1):
- Nottingham University Hospitals NHS Trust, Queens Medical Centre Campus, Nottingham, Nottinghamshire, United Kingdom